CLINICAL TRIAL: NCT04735952
Title: Improving P. Aeruginosa Detection With Breath-based Diagnostics (IMPACT-Breath)
Acronym: IMPACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Arizona State University (Other); Children's Hospital Colorado (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Jane Hill, PhD, Associate Professor, University of British Columbia
Other Study IDs: 331178/ H20-00071; Pro00043176 (Other: Advarra); HILL18A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation); R56HL139846 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-02-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis
Keywords: Breath; IMPACT
MeSH Terms: conditions — Cystic Fibrosis; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breath Samples (The act of analyzing the sample will completely deplete the sample.) Sputum Samples (A portion of the sample may be retained)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIM 1: No-Intervention. Participants in this group will have 1 study visit only. During that visit, breath and sputum samples will be collected.
- AIM 2: No-Intervention. Participants in this group will have up to 8 study visits over a 2 year period. During the study visits, breath and sputum samples will be collected.

SUMMARY:
The study is a breath biomarker validation study. It is anticipated that 300 patients with cystic fibrosis (CF) from 5 clinical sites in the USA will be enrolled. The study is funded by the US NIH and the US Cystic Fibrosis Foundation. Enrollment commenced in May 2019. Sputum, induced sputum, and oropharyngeal swabs will be collected and evaluated at each clinic as part of standard clinical practice. Excess sputum will be sent to Children's Colorado Hospital for molecular analysis. No swabs will be sent anywhere (other than the clinic from which they originate). Breath samples will be taken from all study participants.

DETAILED DESCRIPTION:
AIM 1: Refine and validate volatile biomarkers in the breath of adult and pediatric CF patients for detecting established P. aeruginosa lung infections. For each expectorating subject (n ≥ 288; 5 centers), the diagnostic accuracy of the volatile biomarker panel will be tested, with sputum culture as the standard.

AIM 2: Quantify intra-subject breath variability of the target pediatric population. We will collect longitudinal breath samples for two years from P. aeruginosa-negative subjects (n ≥ 58; ~60% non-expectorating) at 4 pediatric CF clinical centers. We will measure intra-subject variance in the breath signatures of expectorating and non-expectorating subjects, with the latter being the target population for the clinical trial. Two to 8 breath samples will be collected per patient.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1, Cross-Sectional

IInclusion Criteria:

1. Male or female, ages 8 years and older
2. Diagnosis of CF based on sweat chloride ≥ 60 mmol/L and/or 2 known CF mutations
3. @ BC Children's Hospital only- Non-expectorators are eligible if having a clinically indicated OP swab.
4. FEV1 ≥ 30% predicted for spontaneous expectorators or FEV1 ≥ 40% predicted for subjects undergoing sputum induction
5. Either P. aeruginosa (Pa) negative or chronically infected with P. aeruginosa (Pa positive) as defined below:

   a. P. aeruginosa negative: must meet one of the following criteria: i: No growth of Pa in previous 12 months and ≥ 4 consecutive Pa-negative cultures, OR ii: No history of Pa positive airway cultures (sputum, OP, Bronchoalveolar lavage) b. P. aeruginosa positive i: Over 50% of cultures positive and at least 2 cultures positive for Pa in previous 18 months
6. Willing to participate in and comply with the study procedures and willingness of the subject, parent or legally authorized representative to provide written informed consent.

Exclusion criteria:

1. Age < 8 years
2. Intermittently infected with Pa
3. FEV1 < 30%
4. History of lung transplant
5. Presence of a condition or abnormality that in the opinion of the Principal Investigator would compromise the safety of the subject or the quality of the data.

Aim 2, Longitudinal

Inclusion Criteria, Expectorating Cohort (n=48):

1. Male or female, ages 8-16 years
2. Diagnosis of CF based on sweat chloride ≥ 60 mmol/L and/or 2 known CF mutations
3. @ BC Children's Hospital only- Non-expectorators are eligible if having a clinically indicated OP swab.
4. FEV1 ≥ 30% predicted for spontaneous expectorators or FEV1 ≥ 40% predicted for subjects undergoing sputum induction
5. P. aeruginosa negative, based on one of the following criteria:

   1. No growth of Pa in previous 12 months and ≥ 4 consecutive Pa-negative cultures
   2. No history of Pa positive airway cultures (sputum, OP, bronchoalveolar lavage)
6. Willing to participate in and comply with the study procedures and willingness of the subject, parent or legally authorized representative to provide written informed consent.

Exclusion criteria:

1. Age < 8 years
2. Intermittently or chronically infected with Pa
3. Unable to expectorate sputum or undergo sputum induction
4. FEV1 < 30%
5. History of lung transplant
6. Presence of a condition or abnormality that in the opinion of the Principal Investigator would compromise the safety of the subject or the quality of the data.

Inclusion Criteria, Non-Expectorating Cohort (n=10):

1. Male or female, ages 3-8 years
2. Diagnosis of CF based on sweat chloride ≥ 60 mmol/L and/or 2 known CF mutations 3. FEV1 ≥ 30%

4. Unable to expectorate sputum 5. P. aeruginosa negative, based on one of the following criteria:

1. No growth of Pa in previous 12 months and ≥ 4 consecutive Pa-negative cultures
2. No history of Pa positive airway cultures (sputum, OP, bronchoalveolar lavage) 6. Willing to participate in and comply with the study procedures and willingness of the subject, parent or legally authorized representative to provide written informed consent.

Exclusion criteria:

1. Age < 3 years
2. Intermittently or chronically infected with Pa
3. FEV1 < 30%
4. History of lung transplant
5. Presence of a condition or abnormality that in the opinion of the Principal Investigator would compromise the safety of the subject or the quality of the data.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have a diagnosis of cystic fibrosis with cultures that are either P. aeruginosa (Pa) negative or Pa positive.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in concentrations of individual volatile biomarkers and combinations of biomarkers in breath samples obtained from persons with and without P. aeruginosa lung infections | Enrollment thru 2023. Last Longitudinal Study Visit will be 24 months after last AIM 2 enrollment
  Measured using comprehensive two-dimensional gas chromatography of exhaled breath compared to sputum culture (gold standard)

SECONDARY OUTCOMES:
Intra-subject changes in concentrations of individual volatile biomarkers and combinations of biomarkers in breath samples | Thru end of 2025
  Breath samples obtained over a duration of two years, measured using comprehensive two-dimensional gas chromatography of exhaled breath

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Hill, PhD, Principal Investigator — University of British Columbia
Locations (7):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cincinnati Children's Hospital, Cincinnati, Ohio
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Public access to study information and clinical site portal. — http://impactbreath.org